CLINICAL TRIAL: NCT04756349
Title: Clinical Performance of Adhesive Systems Containing HEMA and 10-MDP in Non Carious Cervical Lesions - A Two Years Randomized Double Blind Study
Brief Title: Clinical Performance of Adhesive Systems Containing HEMA and 10-MDP in Non Carious Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Para (Other)
Responsible Party: Principal Investigator, Cecy Martins Silva, Clinical professor, Universidade Federal do Para
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFPara
Record Dates: First submitted 2021-02-05; First posted 2021-02-16 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Non Carious Cervical Lesion
Keywords: adhesives; dental bonding
MeSH Terms: interventions — PRIME protocol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Clearfil SE (Active Comparator): Group containing 10-MDP and HEMA monomers
  Interventions: Other: composite resin restoration
- Optibond All-in-One (Active Comparator): Group containing HEMA monomer
  Interventions: Other: composite resin restoration
- Prime & Bond Universal (Active Comparator): Control Group containing other monomers
  Interventions: Other: composite resin restoration

INTERVENTIONS:
Other: composite resin restoration — All patients will receive adhesive composite resin restorations. There will be 3 groups (different adhesives): Clearfil SE, Optibond All-in-One and Prime & Bond Universal.
  Other Names: composite resin restorations with Clearfil SE adhesive; composite resin restorations with Optibond All-in-One adhesive; composite resin restorations with Prime & Bond Universal adhesive

SUMMARY:
The objective of this randomized, double-blind clinical trial is to evaluate the clinical performance of non-carious cervicals adhesive restorations using three self-etching adhesives containing HEMA and 10-MDP monomers.

DETAILED DESCRIPTION:
Sixty teeth (n = 20 for each group) will be randomized into 03 groups: Clearfil SE (contains MDP and HEMA), Optibond All-inOne (contains HEMA) and Prime and Bond Universal (contains neither monomer) dispatch). Restorations will be performed by a single operator, and no mechanical retention will be performed under the cavity. After 6, 12 and 24 months, the restorations will be evaluated by two calibrated examiners, using modified USPHS criteria for retention (kappa = 1.00) and adaptation / marginal color (kappa = 0.81), and the results will be analysed by Fisher and Kruskal-Wallis, respectively. An intragroup analysis will be performed using the Cochran test (for retention) and Wilcoxon (for marginal adaptation / staining).

ELIGIBILITY:
Inclusion Criteria:

* Good oral hygiene
* Absence of periodontal disease
* Presence of at least 02 non-carious cervical lesions

Exclusion Criteria:

* Presence of non-carious cervical lesion in non-vital teeth
* Occlusal instability
* Presence of orthodontic appliance
* Presence of removable partial dental prosthesis
* High risk of caries (presence of three or more active caries lesions)
* Xerostomia
* Bruxism
* Patients allergic to base materials monomers
* Patients who do not accept the project conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Retention rate of restoration | 01 year
  The retention rate will be assessed following the USPHS (United States Public Health) guidelines with the following classifications (acronyms):
  Alpha = retained. Charlie = mobility or loss.
Retention rate of restoration | 02 years
  The retention rate will be assessed following the USPHS (United States Public Health) guidelines with the following classifications (acronyms):
  Alpha = retained. Charlie = mobility or loss.

SECONDARY OUTCOMES:
Marginal staining rate of restoration | 01 year
  The marginal staining rate will be assessed following the USPHS (United States Public Health) guidelines with the following classifications (acronyms):
  Alpha = no staining. Bravo = superficial staining (localized or generalized). Charlie = deep staining (localized or generalized).
Marginal staining rate of restoration | 02 years
  The marginal staining rate will be assessed following the USPHS (United States Public Health) guidelines with the following classifications (acronyms):
  Alpha = no staining. Bravo = superficial staining (localized or generalized). Charlie = deep staining (localized or generalized).
Marginal Adaptation rate of restoration | 01 year
  The marginal adaptation rate will be assessed following the USPHS (United States Public Health) guidelines with the following classifications (acronyms):
  Alpha = no visible evidence of a crack along the edge, the explorer will not penetrate.
  Bravo = visible evidence of a crack along the margin, dentin unexposed, clinically acceptable.
  Charlie = explorer penetrates the crack, dentin exposed, clinically unacceptable.
Marginal Adaptation rate of restoration | 02 years
  The marginal adaptation rate will be assessed following the USPHS (United States Public Health) guidelines with the following classifications (acronyms):
  Alpha = no visible evidence of a crack along the edge, the explorer will not penetrate.
  Bravo = visible evidence of a crack along the margin, dentin unexposed, clinically acceptable.
  Charlie = explorer penetrates the crack, dentin exposed, clinically unacceptable.

OTHER OUTCOMES:
Postoperative sensitivity rate of restoration | 01 year
  present or absent
Postoperative sensitivity rate of restoration | 02 years
  present or absent
Secondary caries rate of restoration | 01 year
  present or absent
Secondary caries rate of restoration | 02 years
  present or absent

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Oliveira, Msc, Principal Investigator — Federal University of Pará; Brennda De Paula, Msc, Study Chair — Federal University of Pará; Cecy Silva, PhD, Study Director — Federal University of Pará
Locations (1):
- Para's Federal University, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: No